CLINICAL TRIAL: NCT00005954
Title: Phase II Treatment of Adults With Brain Metastases With Temodar
Brief Title: Temozolomide in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Henry Friedman, MD, Duke UMC
Purpose: Treatment
Other Study IDs: 2114; DUMC-2114-02-12R3; NCI-G00-1798; CDR0000067934 (Other: NCI)
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult tumors metastatic to brain
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of temozolomide in treating patients who have brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the activity of temozolomide in patients with brain metastases.
* Determine the toxicity of this treatment in these patients.

OUTLINE: Patients are stratified according to type of primary cancer (lung carcinoma vs breast carcinoma vs malignant melanoma vs renal cell carcinoma vs colorectal carcinoma vs other).

Patients receive oral temozolomide daily on days 1-7 and 15-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 180 patients (30 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Metastatic lesions to the brain

  * Must not require immediate radiotherapy
  * If received prior radiotherapy, must have progressive disease
* Evaluable disease by CT scan or MRI
* Neurologically stable

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* SGOT or SGPT less than 2.5 times ULN
* Alkaline phosphatase less than 2 times ULN

Renal:

* Blood urea nitrogen less than 1.5 times ULN
* Creatinine less than 1.5 times ULN

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other concurrent nonmalignant systemic disease
* No acute infection requiring treatment with IV antibiotics
* HIV negative
* No frequent vomiting or medical condition that would preclude oral medication administration (e.g., partial bowel obstruction, inability to swallow)

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent hematopoietic growth factors, including epoetin alfa
* No other concurrent biologic therapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy, unless evidence of disease progression
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent corticosteroids allowed if nonincreasing dose for at least 1 week prior to study

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy to the brain, unless evidence of disease progression
* No concurrent radiotherapy

Surgery:

* At least 3 weeks since prior surgery, unless evidence of disease progression, and recovered

Other:

* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08; Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States